CLINICAL TRIAL: NCT00812968
Title: A Multicenter, Single-arm Study to Assess the Safety, Pharmacokinetics and Efficacy of Lenalidomide in Japanese Subjects With Low- or Intern=Mediate-1-risk Myelodysplastic Syndromes (MDS) Associated With a Deletion 5 (q31-33) Abnormality and Symptomatic Anemia
Brief Title: Study of CC-5013 to Evaluate Safety, Pharmacokinetics and Effectiveness for Japanese Patients With Symptomatic Anemia Associated With Myelodysplastic Syndrome With a Del(5)(q31-33) Abnormality.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-MDS-007
Record Dates: First submitted 2008-12-17; First posted 2008-12-22 (Estimated); Results first posted 2013-12-17 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic Syndromes; Lenalidomide
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental): Oral 10mg daily on Days 1-21 days every 28 days until disease progression/relapse or CC-5013 is permanently discontinued for any reason for up to 156 weeks (3 years).
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Oral 10mg daily on Days 1-21 days every 28 days until disease progression/relapse or CC-5013 is permanently discontinued for any reason for up to 156 weeks (3 years).
  Other Names: CC-5013

SUMMARY:
The purpose of this clinical experience study is to determine whether CC-5013 is safe and effective (to include studying the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body [pharmacokinetics]) in Japanese subjects with low- or intermediate-1-risk MDS (IPSS risk categories) associated with a deletion 5(q31-33) abnormality and symptomatic anemia.

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign an informed consent form.
* Age ≥ 20 years at the time of signing the informed consent form.
* Must be able to adhere to the study visit schedule and other protocol requirements.
* Diagnosis of Myelodysplastic Syndrome (MDS) that meets International Prognostic Scoring System (IPSS) criteria for low- or intermediate-1-risk disease associated with a deletion 5(q31-33) abnormality
* Symptomatic anemia secondary to MDS defined as:Untransfused Hb level < 10.0 g/dL and a Functional Assessment of Cancer Therapy (FACT)-anemia subscale score of ≤ 74 or Transfusion dependent anemia

Exclusion Criteria:

* Pregnant or lactating females.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
* Prior therapy with lenalidomide.
* Patients with any of the following laboratory abnormalities within 14 days of starting study drug: Absolute Neutrophil Count (ANC) < 750 cells/μL (0.75 x 10^9/L) Platelet count < 50,000/μL (50x10^9/L) Serum creatinine > 2.5 mg/dL Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) > 3.0 x Upper Limit of Normal (ULN)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-09-01 (Actual); Primary Completion 2010-09-01 (Actual); Study Completion 2010-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masaaki Takatoku, MD, Study Director — Celgene Corporation
Locations (6):
- Japan (6):
  - Celgene Clinical Site, Shimono, Tochigi
  - Celgene Clinical Site, Shibuya-ku, Tokyo
  - Celgene Clinical Site, Hiroshima
  - Celgene Clinical Site, Kyoto
  - Celgene Clinical Site, Osaka
  - Celgene Clinical Site, Shizuoka

REFERENCES:
- [Background] Matsuda A, Taniwaki M, Jinnai I, Harada H, Watanabe M, Suzuki K, Yanagita S, Suzuki T, Yoshida Y, Kimura A, Tsudo M, Tohyama K, Takatoku M, Ozawa K. Morphologic analysis in myelodysplastic syndromes with del(5q) treated with lenalidomide. A Japanese multiinstitutional study. Leuk Res. 2012 May;36(5):575-80. doi: 10.1016/j.leukres.2011.11.011. Epub 2011 Dec 15. PMID 22172461
- [Result] Harada H, Watanabe M, Suzuki K, Yanagita S, Suzuki T, Yoshida Y, Kimura A, Tsudo M, Matsuda A, Tohyama K, Taniwaki M, Takeshita K, Takatoku M, Ozawa K. Lenalidomide is active in Japanese patients with symptomatic anemia in low- or intermediate-1 risk myelodysplastic syndromes with a deletion 5q abnormality. Int J Hematol. 2009 Oct;90(3):353-360. doi: 10.1007/s12185-009-0400-8. Epub 2009 Aug 25. PMID 19705057

RESULTS

PARTICIPANT FLOW:
Groups:
- Lenalidomide: 10 mg of lenalidomide was administered orally once daily on Days 1 to 21 of every 28-day cycle. Treatment continued until disease progression or relapse following an erythroid improvement was documented, any of the criteria for treatment discontinuation was violated, or lenalidomide became commercially available for the treatment of MDS associated with a del (5q) cytogenetic abnormality, for up to 156 weeks (3 years).
Period: Overall Study
Arm/Group | Lenalidomide
Started | 11
Completed | 0
Not Completed | 11
Not completed — Relapse after erythroid response | 6
Not completed — Disease progression | 1
Not completed — No further treatment required | 1
Not completed — Study closed due to marketing approval | 3

BASELINE CHARACTERISTICS:
Groups:
- Lenalidomide: 10 mg of lenalidomide was administered orally once daily on Days 1 to 21 of every 28-day cycle, for up to 156 weeks (3 years).
Arm/Group | Lenalidomide
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.8 (5.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Region of Enrollment [Number; unit: participants]
  Japan | 11
Duration of MDS [Mean (Standard Deviation); unit: years] | 2.0 (1.44)
International Prognostic Scoring System (IPSS) Score [Number; unit: participants] — The MDS IPSS assesses the severity of MDS based on 3 prognostic factors each assigned a score: the proportion of bone marrow blasts, chromosome changes in the marrow cells (karyotype) and the presence of one or more low blood cell counts (cytopenias). The IPSS score is the sum of the bone marrow blast + karyotype + cytopenia score and ranges from 0 (low risk) to 3.5 (high risk). Prognosis is categorized as Low risk (score = 0), Intermediate-1 (score 0.5 to 1.0), Intermediate-2 (score 1.5 to 2.0) or High risk (score ≥ 2.5).
  participants
    Low risk | 2
    Intermediate-1 risk | 9
    Intermediate-2 risk | 0
    High risk | 0
French-American-British (FAB) classification of MDS [Number; unit: participants] — The French-American-British (FAB) classification of MDS recognizes five subtypes of MDS that are distinguished by the percentage of myeloblasts, presence or absence of ringed sideroblasts (i.e., erythroid precursors with iron deposits surrounding the nucleus), or a monocytosis.
  participants
    Refractory anemia (RA) | 9
    Refractory anemia with ringed sideroblasts (RARS) | 0
    Refractory anemia with excess blasts (RAEB) | 2
    Chronic myelomonocytic leukemia (CMML) | 0
    RAEB in transformation (RAEB-t) | 0
World Health Organization Classification of MDS [Number; unit: participants] — The World Health Organization (WHO) classification recognizes eight subtypes of MDS that are distinguished by the percentage of myeloblasts, presence or absence of ringed sideroblasts (i.e., erythroid precursors with iron deposits surrounding the nucleus), presence of a monocytosis or a deletion 5q.
  participants
    Refractory anemia (RA) | 0
    RA with ringed sideroblasts (RARS) | 0
    Refractory anemia with excess blasts-1 (RAEB-1) | 2
    Refractory anemia with excess blasts-2 (RAEB-2) | 0
    Refractory cytopenia multilineage dysplasia (RCMD) | 1
    RCMD and ringed sideroblasts (RCMD-RS) | 0
    MDS, unclassified (MDS-U) | 0
    MDS associated with isolated del(5q) | 8
Bone Marrow Cellularity [Number; unit: participants] — Bone marrow cellularity is a measure of the percentage of hematopoietic stem cells relative to fat cells in the bone marrow.
  participants
    Aplastic (0%) | 0
    Hypocellular (> 0% to ≤ 30%) | 3
    Normocellular (> 30% to ≤ 60%) | 5
    Hypercellular (> 60% to ≤ 90%) | 2
    Packed (> 90% to ≤ 100%) | 0
    Missing | 1
Transfusion Dependency [Number; unit: participants]
  Yes | 5
  No | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AE)
Description: An AE that resulted in any of the following outcomes was defined as a serious adverse event (SAE):
  * Death;
  * Life-threatening event;
  * Any inpatient hospitalization or prolongation of existing hospitalization;
  * Persistent or significant disability or incapacity;
  * Congenital anomaly or birth defect;
  * Any other important medical event.
  The investigator determined the relationship of an AE to study drug based on the timing of the AE relative to drug administration and whether or not other drugs, therapeutic interventions, or underlying conditions could provide a sufficient explanation for the event.
  The severity of an AE was evaluated by the investigator according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (Version 3.0) where Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Life-threatening and Grade 5 = Death.
Time Frame: After the first study dose until 28 days after completion of/discontinuation from the study (maximum time on study was 155 weeks).
Population: Safety population: all patients who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 11
participants
  Any adverse event (AE) | 11
  AE related to study drug | 11
  Grade 3 or 4 AE | 11
  Grade 3 or 4 AE related to study drug | 11
  Serious AE (SAE) | 3
  SAE related to study drug | 1
  AE leading to discontinuation of study drug | 0
  Related AE leading to discontinuation | 0
  AE leading to a dose reduction or interruption | 10
  Related AE leading to dose reduction/interruption | 9
  Deaths | 0

2. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Lenalidomide
Description: Maximum observed plasma concentration of lenalidomide after a single dose on Day and after multiple doses (Day 4).
Time Frame: Days 1 and 4 at predose and 0.5, 1, 1.5, 2, 3, 4, 6, 9, and 12 hours post-dose.
Population: Pharmacokinetic (PK) population: all patients who adhered to the study treatment during the course of PK assessment (Days 1 to 5 of Cycle 1) and from whom blood and urine samples were collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Lenalidomide: Day 1: Analysis of PK parameters on Day 1, after a single dose of 10 mg of lenalidomide administered orally.
- Lenalidomide: Day 4: Analysis of PK parameters on Day 4, after participants had received 10 mg of lenalidomide administered orally once daily for 4 days.
Arm/Group | Lenalidomide: Day 1 | Lenalidomide: Day 4
Number analyzed (Participants) | 6 | 5
ng/mL | 136 (43.1) | 149 (31.2)

3. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Lenalidomide
Description: Time to maximum observed plasma concentration of lenalidomide after a single dose on Day 1 and multiple doses (Day 4).
Time Frame: Days 1 and 4 at predose and 0.5, 1, 1.5, 2, 3, 4, 6, 9, and 12 hours post-dose.
Population: PK population
Measure: Median (Full Range); unit: hours
Arm/Group | Lenalidomide: Day 1 | Lenalidomide: Day 4
Number analyzed (Participants) | 6 | 5
hours | 2.52 [1.00 to 5.95] | 2.93 [1.00 to 4.00]

4. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Measurable Concentration (AUCt) of Lenalidomide
Description: Area under the plasma concentration-time curve from time zero to the last measurable concentration (AUCt) of lenalidomide after a single dose on Day 1 and multiple doses (Day 4).
Time Frame: Days 1 and 4 at predose and 0.5, 1, 1.5, 2, 3, 4, 6, 9, and 12 hours post-dose.
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Lenalidomide: Day 1 | Lenalidomide: Day 4
Number analyzed (Participants) | 6 | 5
ng*h/mL | 718.4 (41.2) | 803.5 (46.9)

5. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over the Dosing Interval (AUCτ) of Lenalidomide
Description: Area under the plasma concentration-time curve over the dosing interval (AUCτ) of lenalidomide after a single dose on Day 1 and multiple doses (Day 4).
Time Frame: Days 1 and 4 at predose and 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12 and 24 hours post-dose.
Population: PK population with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Lenalidomide: Day 1 | Lenalidomide: Day 4
Number analyzed (Participants) | 5 | 5
ng*h/mL | 866.5 (44.1) | 877.9 (43.0)

6. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC∞) of Lenalidomide
Description: Area under the plasma concentration-time curve from time zero to infinity (AUC∞) of lenalidomide after a single dose on Day 1.
Time Frame: Day 1 at predose and 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12 and 24 hours post-dose.
Population: PK population with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Lenalidomide
Number analyzed (Participants) | 5
ng*h/mL | 878.0 (45.1)

7. Secondary Outcome: Terminal Half-life (T1/2) of Lenalidomide
Description: The apparent terminal half-life is the time required for plasma concentration to decrease by 50% after pseudo-equilibrium of distribution has been reached, and calculated as the natural logarithm of 2 (0.693) / Apparent terminal rate constant (λz).
Time Frame: Days 1 and 4 at predose and 0.5, 1, 1.5, 2, 3, 4, 6, 9, and 12 hours post-dose.
Population: PK population with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Lenalidomide: Day 1 | Lenalidomide: Day 4
Number analyzed (Participants) | 5 | 5
hours | 3.26 (23.0) | 3.57 (29.6)

8. Secondary Outcome: Apparent Volume of Distribution (VzF) of Lenalidomide
Description: Apparent volume of distribution of lenalidomide after a single dose on Day 1 and multiple doses (Day 4).
Time Frame: Days 1 and 4 at predose and 0.5, 1, 1.5, 2, 3, 4, 6, 9, and 12 hours post-dose.
Population: PK population with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Lenalidomide: Day 1 | Lenalidomide: Day 4
Number analyzed (Participants) | 5 | 5
liters | 53.6 (30.9) | 58.6 (25.8)

9. Secondary Outcome: Apparent Total Plasma Clearance (CL/F) of Lenalidomide
Description: Apparent total plasma clearance (CL/F) of lenalidomide after a single dose on Day 1 and multiple doses (Day 4).
Time Frame: Days 1 and 4 at predose and 0.5, 1, 1.5, 2, 3, 4, 6, 9, and 12 hours post-dose.
Population: PK population with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/minute
Arm/Group | Lenalidomide: Day 1 | Lenalidomide: Day 4
Number analyzed (Participants) | 5 | 5
mL/minute | 189.8 (45.1) | 189.9 (43.0)

10. Secondary Outcome: Apparent Terminal Elimination Rate Constant of Lenalidomide
Description: Apparent terminal elimination rate constant of lenalidomide determined after a single dose on Day 1 and multiple doses (Day 4).
Time Frame: Days 1 and 4 at predose and 0.5, 1, 1.5, 2, 3, 4, 6, 9, and 12 hours post-dose.
Population: PK population with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Lenalidomide: Day 1 | Lenalidomide: Day 4
Number analyzed (Participants) | 5 | 5
1/h | 0.213 (23.0) | 0.194 (39.0)

11. Secondary Outcome: Number of Participants With a Erythroid Response
Description: Erythroid response was determined using the International Working Group (IWG) 2000 criteria, categorized as a major response or minor response.
  A major response in patients with transfusion-dependent anemia (receiving ≥ 4.5 units of red blood cell (RBC) transfusion during 56 consecutive days at Baseline) is defined as RBC transfusion independence accompanied by a ≥1.0 g/dL increase from Baseline in hemoglobin sustained for 56 days consecutively during the treatment period. In patients with transfusion-independent anemia with hemoglobin < 10 g/dL at Baseline a major response is defined as a > 2.0 g/dL increase from Baseline in hemoglobin sustained for consecutive 56 days.
  Minor response in patients with transfusion-dependent anemia defined as ≥ 50% decrease from Baseline in transfusion requirements sustained for consecutive 56 days, and in transfusion-independent patients as 1.0 to 2.0 g/dL increase from Baseline in hemoglobin sustained for consecutive 56 days.
Time Frame: Response was assessed every 28 days through Week 156.
Population: Efficacy population: all patients who had a diagnosis of low- or intermediate-1-risk MDS associated with anemia based on confirmation by the central reviewers and received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 11
participants
  Erythroid responders (major or minor) | 11
  Major erythroid responders | 11

12. Secondary Outcome: Time to Erythroid Response
Description: Time to erythroid response was calculated as the time from the first dose of study drug to the start of the first major or minor erythroid response. Similarly, time to major erythroid response was calculated as the time from the first dose of study drug to the start of the first major erythroid response.
Time Frame: From the first dose of study drug through Week 156
Population: Efficacy population
Measure: Median (Full Range); unit: weeks
Arm/Group | Lenalidomide
Number analyzed (Participants) | 11
weeks
  Time to erythroid response (major or minor) | 2.1 [0.3 to 11.1]
  Time to major erythroid response | 6.3 [3.1 to 31.1]

13. Secondary Outcome: Duration of Erythroid Response
Description: Duration of erythroid response was calculated as the time from the start of the first major or minor erythroid response to the end of the response. Similarly, duration of major erythroid response was calculated as the time from the start of the first major erythroid response to the end of the response. Response duration was censored at the last adequate assessment for patients who maintained response.
Time Frame: From the first dose of study drug through Week 156
Population: Efficacy population with a erythroid response
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenalidomide
Number analyzed (Participants) | 11
weeks
  Duration of erythroid response (major or minor) | 76.6 [8.9 to 152.0]
  Duration of major erythroid response | 72.1 [32.1 to 144.1]

14. Secondary Outcome: Change From Baseline in Hemoglobin Concentration
Description: Change in hemoglobin concentration from Baseline to the maximum observed value during the major erythroid response period for major erythroid responders.
Time Frame: Baseline and from Day1 until the maximum observed value (up to 155 weeks)
Population: Efficacy population with a erythroid response
Measure: Median (Full Range); unit: g/dL
Arm/Group | Lenalidomide
Number analyzed (Participants) | 11
g/dL
  Baseline concentration | 7.0 [4.7 to 9.1]
  Maximum concentration during study | 13.1 [10.7 to 15.8]
  Change from Baseline to maximum value | 6.0 [2.7 to 11.1]

15. Secondary Outcome: Number of Participants With a Neutrophil Response
Description: Neutrophil response was determined using the IWG (2000) criteria. A major response for participants with a Baseline neutrophil count < 1,500/mm^3 is defined as a ≥ 100% increase or a ≥ 500/mm^3 increase, whichever is greater, sustained for consecutive 56 days during the treatment period.
  A minor response for participants with a Baseline neutrophil count < 1,500/mm^3 is defined as a ≥ 100% increase, but an absolute increase < 500/mm^3, sustained for consecutive 56 days during the treatment period.
Time Frame: Response was assessed every 28 days through Week 156
Population: Efficacy population with Baseline neutrophil count < 1,500/mm^3.
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 6
participants
  Major response | 1
  Minor response | 0

16. Secondary Outcome: Number of Participants With a Platelet Response
Description: Platelet response was determined using the IWG (2000) criteria. Major response in patients with Baseline platelet count < 100,000/mm^3 is defined as a ≥ 30,000/mm^3 increase sustained for consecutive 56 days during the treatment period. In platelet-transfusion-dependent patients at Baseline a major response is defined as stabilization of platelet counts and platelet transfusion independence sustained for consecutive 56 days during the treatment period.
  Minor response in patients with Baseline platelet count < 100,000/mm^3 is defined as a ≥ 50% increase in platelet count with an absolute increase > 10,000/mm^3 and < 30,000/mm^3 sustained for consecutive 56 days during the treatment period.
Time Frame: Response was assessed every 28 days through Week 156
Population: Efficacy population with a Baseline platelet count of < 100,000/mm^3 or who were platelet-transfusion dependent at Baseline. There were no patients with platelet count of < 100,000/mm3 or who were platelet-transfusion dependent at Baseline, and thus platelet response was not evaluated.
Arm/Group | Lenalidomide
Number analyzed (Participants) | 0

17. Secondary Outcome: Number of Participants With a Cytogenetic Response
Description: Cytogenetic (chromosome structure) abnormalities were assessed by a central cytogenetic reviewer based on prints and cytogenetic reports of the bone marrow sample from the central laboratory. Cytogenetic response was determined using the IWG (2000) criteria and categorized as either a major response or minor response. Twenty metaphases were analyzed for the determination of cytogenetic response.
  A major response was defined as no detectable cytogenetic abnormality, if an abnormality was present at Baseline, sustained for consecutive 56 days during the treatment period. A minor response was defined as ≥ 50% reduction from Baseline in abnormal metaphases sustained for consecutive 56 days during the treatment period.
Time Frame: Response was assessed every 12 weeks through Week 156
Population: Efficacy population
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 11
participants
  Major response | 1
  Minor response | 5

18. Secondary Outcome: Change From Baseline in Percentage of Bone Marrow Erythroblasts
Description: Bone marrow morphology was assessed by the central hematologic reviewers based on the locally-prepared bone marrow smear slide and clot section.
Time Frame: Baseline, at the end of Cycle 3 (Day 85) and Cycle 6 (Day 169).
Population: Efficacy population with available bone marrow specimens.
Measure: Median (Full Range); unit: Percentage of Bone Marrow Erythroblasts
Arm/Group | Lenalidomide
Number analyzed (Participants) | 10
Percentage of Bone Marrow Erythroblasts
  Change from Baseline at the end of Cycle 3 | 36.5 [-12.0 to 51.0]
  Change from Baseline at the end of Cycle 6 | 21.5 [-5.0 to 56.0]

19. Secondary Outcome: Percentage of Bone Marrow Myeloblasts
Description: as for outcome 18
Time Frame: Baseline, at the end of Cycle 3 (Day 85) and Cycle 6 (Day 169).
Population: Efficacy population with available bone marrow specimens at each time point (indicated by "N").
Measure: Median (Full Range); unit: Percentage of myeloblasts
Arm/Group | Lenalidomide
Number analyzed (Participants) | 11
Percentage of myeloblasts
  Baseline (N=11) | 3.77 [1.20 to 8.40]
  End of Cycle 3 (N=10) | 1.47 [0.01 to 4.55]
  End of Cycle 6 (N=10) | 1.79 [0.01 to 4.00]

20. Secondary Outcome: Percentage of Bone Marrow Promyelocytes
Description: as for outcome 18
Time Frame: Baseline, at the end of Cycle 3 (Day 85) and Cycle 6 (Day 169).
Population: Efficacy population with available bone marrow specimens at each time point (indicated by "N").
Measure: Median (Full Range); unit: Percentage of promyelocytes
Arm/Group | Lenalidomide
Number analyzed (Participants) | 11
Percentage of promyelocytes
  Baseline (N=11) | 5 [0 to 13]
  End of Cycle 3 (N=10) | 5 [1 to 12]
  End of Cycle 6 (N=10) | 5 [1 to 12]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug through 28 days after completion of/discontinuation from the study (maximum time on study was 155 weeks).
Arm/Group | Lenalidomide
Serious Adverse Events (participants affected / at risk) | 3/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=11)
Gastric Ulcer (Gastrointestinal disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Herpes Zoster (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1
Liver Function Test Abnormal (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=11)
Neutropenia (Blood and lymphatic system disorders) | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 11
Leukopenia (Blood and lymphatic system disorders) | 10
Lymphopenia (Blood and lymphatic system disorders) | 8
Eosinophilia (Blood and lymphatic system disorders) | 5
Basophilia (Blood and lymphatic system disorders) | 4
Leukocytosis (Blood and lymphatic system disorders) | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1
Lymphocytosis (Blood and lymphatic system disorders) | 1
Constipation (Gastrointestinal disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 4
Abdominal Pain (Gastrointestinal disorders) | 2
Dental Caries (Gastrointestinal disorders) | 2
Enteritis (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 2
Abdominal Discomfort (Gastrointestinal disorders) | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Dyspepsia (General disorders) | 1
Gingivitis (Gastrointestinal disorders) | 1
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1
Lip Dry (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Periodontitis (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Nasopharyngitis (Infections and infestations) | 8
Bronchitis (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 3
Rhinitis (Infections and infestations) | 2
Urinary Tract Infection (Infections and infestations) | 2
Acute Tonsillitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Lymphadenitis Bacterial (Infections and infestations) | 1
Oral Herpes (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Vulvitis (Infections and infestations) | 1
Rash (Skin and subcutaneous tissue disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 5
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 4
Eczema (Skin and subcutaneous tissue disorders) | 2
Acute Febrile Neutrophilic Dermatosis (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1
Alanine Aminotransferase Increased (Investigations) | 3
Blood Creatinine Increased (Investigations) | 3
Fibrin Degradation Products Increased (Investigations) | 3
Aspartate Aminotransferase Increased (Investigations) | 2
Blood Bilirubin Increased (Investigations) | 2
Blood Phosphorus Decreased (Investigations) | 2
Blood Uric Acid Increased (Investigations) | 2
Fibrin D Dimer Increased (Investigations) | 2
Blood Alkaline Phosphatase Increased (Investigations) | 1
Blood Lactate Dehydrogenase Increased (Investigations) | 1
Blood Potassium Increased (Investigations) | 1
Blood Pressure Increased (Investigations) | 1
Blood Urea Decreased (Investigations) | 1
Blood Urea Increased (Investigations) | 1
International Normalised Ratio Increased (Investigations) | 1
Mean Cell Volume Increased (Investigations) | 1
Protein Total Increased (Investigations) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 4
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Myalgia Intercostal (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 3
Contusion (Injury, poisoning and procedural complications) | 3
Excoriation (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Tooth Fracture (Injury, poisoning and procedural complications) | 1
Face Oedema (General disorders) | 1
Injection Site Erythema (General disorders) | 1
Non-cardiac Chest Pain (General disorders) | 1
Oedema (General disorders) | 1
Oedema Peripheral (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Iron Deficiency (Metabolism and nutrition disorders) | 1
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 4
Blepharitis (Eye disorders) | 1
Conjunctival Haemorrhage (Eye disorders) | 1
Eye Discharge (Eye disorders) | 1
Vision Blurred (Eye disorders) | 1
Vitreous Detachment (Eye disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Cervicobrachial Syndrome (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Tension (Psychiatric disorders) | 1
Ear Discomfort (Ear and labyrinth disorders) | 1
Hepatic Function Abnormal (Hepatobiliary disorders) | 1
Dysuria (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure agreements vary; the Investigators shall not disclose any material/information disclosed by the Sponsor (Celgene KK) with the clinical trial or information obtained by conducting the clinical trial to third parties without Sponsor's prior written approval.